CLINICAL TRIAL: NCT00857467
Title: Randomised, Double-blind, Single Dose, Three-way, Cross-over Study to Investigate the Safety and Response to 1g or 2g Rectal Suppositories Containing 5 mg or 10 mg 1R,2S-methoxamine Hydrochloride [NRL001] or Matching Placebo
Brief Title: Study to Investigate Safety and Response to 1 or 2 g Rectal Suppositories Containing 5 or 10 mg NRL001.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Norgine (Industry)
Responsible Party: Vice President Clinical Development, Norgine
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: NRL001-01/2008 (SUM)
Record Dates: First submitted 2009-03-05; First posted 2009-03-06 (Estimated); Last update posted 2009-12-23 (Estimated); Status verified 2009-12

CONDITIONS: Fecal Incontinence
MeSH Terms: conditions — Fecal Incontinence

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 g suppository (Experimental): Subjects receive 5 mg NRL001, 10 mg NRL001 and placebo in a 1g rectal suppository
  Interventions: Drug: NRL001
- 2 g suppository (Experimental): Subjects receive 5 mg NRL001, 10 mg NRL001 and placebo in a 2 g rectal suppository.
  Interventions: Drug: NRL001

INTERVENTIONS:
Drug: NRL001 — Subjects receive single doses of 5 mg NRL001, 10 mg NRL001 and placebo in a 1 g rectal suppository, with a 7-day washout period between dosing.
  Arms: 1 g suppository
Drug: NRL001 — Subjects receive single doses of 5 mg NRL001, 10 mg NRL001 and placebo in a 2 g rectal suppository, with a 7-day washout period between dosing.
  Arms: 2 g suppository

SUMMARY:
This is a healthy volunteer three-way crossover study. A total of 12 subjects will receive three single administrations of 1 g rectal suppositories (containing either 5 mg NRL001, 10 mg NRL001 or matching placebo), with a washout period of at least 7 days between dosings. A further 12 subjects will receive three single administrations of 2 g rectal suppositories (containing either 5 mg NRL001, 10 mg NRL001 or matching placebo), again with a 7 day washout period between dosings. The pharmacodynamic response, pharmacokinetics and safety profile will be determined.

ELIGIBILITY:
Inclusion Criteria:

1. No previous history of ano-rectal conditions or diseases
2. No history of cardiovascular disease
3. 18 to 60 years of age
4. Males and females (pre-menopausal females of child-bearing potential must be using adequate contraceptive methods and have a negative pregnancy test before the start of the study)

Exclusion Criteria:

1. Use of medication in the last 30 days with a vasodilatory activity, or use of any medication currently or within the last 30 days which the Investigator believes may affect the study participation or results
2. Use of monoamine oxidase inhibitors presently or within the last 2 weeks before study participation
3. Use of any medication in the last 30 days applied to the anus and/or via the rectum
4. Application of any unlicensed medication within the previous 3 months or participation in any other research study in the last three months which involved being paid a disturbance allowance; having an invasive procedure (e.g. venepuncture >50ml, endoscopy) or exposure to ionising radiation.
5. Regular intake of more than 21 units of alcohol per week
6. History or any evidence of cardiovascular disease including ischaemic heart disease and hypertension (defined on examination: systolic blood pressure greater than 160 mmHg or diastolic blood pressure greater than 90 mmHg; based on at least two separate readings), peripheral vascular disease or Raynaud's syndrome
7. Presence of diabetes mellitus
8. History or symptoms of thyroid diseases, including hypo- or hyperthyroidism
9. Pregnant or lactating females
10. History of any clinically relevant allergy
11. Presence of concomitant gastrointestinal diseases or disorders, such as significant abdominal symptoms and haemorrhoids but also any significant organ (e.g. renal, hepatic or cardiac) dysfunction
12. Volunteers whom the Investigator feels would not comply with the requirements of the trial
13. Volunteers who have been exposed to more than 5 mSv of ionising radiation in the last 12 months.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2009-02; Primary Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Change in MARP after a single dose | 6 hours

SECONDARY OUTCOMES:
Pharmacokinetic plasma assessment to determine systemic uptake | 6 hours
Adverse events | 6 hours
Cardiovascular parameters; heart rate and blood pressure | 6 hours

CONTACTS AND LOCATIONS:
Overall Officials: Hans-Jürgen Gruss, MD, Study Director — Norgine; John H Scholefield, MD, Principal Investigator — Nottingham University Hospital
Locations (1):
- Department of GI Surgery, Nottingham University Hospital, Nottingham, United Kingdom

REFERENCES:
- [Derived] Simpson JA, Bush D, Gruss HJ, Jacobs A, Pediconi C, Scholefield JH. A randomised, controlled, crossover study to investigate the safety and response of 1R,2S-methoxamine hydrochloride (NRL001) on anal function in healthy volunteers. Colorectal Dis. 2014 Mar;16 Suppl 1:5-15. doi: 10.1111/codi.12541. PMID 24499492